CLINICAL TRIAL: NCT00631306
Title: Effects of Cranberry Juice on Risk Factors for Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Ocean Spray, Inc. (Industry)
Responsible Party: Amir Lerman, MD, Mayo Clinic
Other Study IDs: 07-003443
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bottle number 615: Patients are randomized to either Bottle number 615 or Bottle number 429 (actual product vs. placebo). This is a blinded study.
- Bottle number 429: Patients are randomized to either Bottle number 615 or Bottle number 429 (actual product vs. placebo). This is a blinded study.

SUMMARY:
This study is being done to determine if the use of double strength cranberry juice in daily diet will improve endothelial function.

DETAILED DESCRIPTION:
Study participants will be randomized assigned to drink either placebo (a drink that looks and tastes like cranberry juice, but does not contain cranberry juice) or a double strength Ocean Spray light cranberry juice cocktail for four months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 18 years old with known or suspected cardiovascular disease including documented CAD by cardiac catheterization, and multiple cardiovascular risk factors will be included, regardless of severity of endothelial dysfunction or previous history of cardiovascular events.
* Subjects with no known history of cardiac disease will also be eligible to participate.
* Subjects must demonstrate endothelial dysfunction via the RH-PAT test (an RH-PAT score of less than 2.0) to continue participating in this study.

Exclusion Criteria:

* Patients will be excluded if they have confounding factors including, but not limited to, history of renal or liver failure, or relevant food allergies (cranberries, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic Patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The current study was designed to test the hypothesis that the chronic administration of supplementation with double-strength cranberry juice will improve peripheral endothelial dysfunction. | baseline and 4 months post

SECONDARY OUTCOMES:
The current study was also designed to test the acute effect of double-strength cranberry juice on endothelial function. | 45 mins post consumption

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Flammer AJ, Martin EA, Gossl M, Widmer RJ, Lennon RJ, Sexton JA, Loeffler D, Khosla S, Lerman LO, Lerman A. Polyphenol-rich cranberry juice has a neutral effect on endothelial function but decreases the fraction of osteocalcin-expressing endothelial progenitor cells. Eur J Nutr. 2013 Feb;52(1):289-96. doi: 10.1007/s00394-012-0334-4. Epub 2012 Mar 2. PMID 22382203